CLINICAL TRIAL: NCT03782142
Title: What is the Impact of Current HIV Medication Regimens on Endothelial Dysfunction?
Brief Title: Effect on HIV Medications on EPC Cells
Status: Completed | Type: Observational
Sponsor: Sabyasachi Sen (Other)
Responsible Party: Sponsor-Investigator, Sabyasachi Sen, Associate Professor, Dept. of Medicine (Division of Endocrinology), George Washington University
Organization: George Washington University (Other)
Other Study IDs: 180510
Record Dates: First submitted 2018-10-17; First posted 2018-12-20 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Rilpivirine; cobicistat mixture with darunavir; dolutegravir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Group A NRTI + NNRTI: Based on current regimens that are commonly used (2017-2018 ART guidelines), our groups will include NRTI such as TAF (tenofovir alafenamide) or TDF (tenofovir disoproxil fumarate) and an NNRTI (Non-nucleoside reverse transcriptase inhibitor, Rilpivirine
  Interventions: Drug: Tenofovir; Drug: Rilpivirine
- Group B NRTI + boosted PI: NRTI such as TAF (tenofovir alafenamide) or TDF (tenofovir disoproxil fumarate) and a boosted Protease Inhibitor: Prezcobix- [darunavir+cobicistat combination]
  Interventions: Drug: Tenofovir; Drug: Prezcobix
- Group C NRTI + II: NRTI such as TAF (tenofovir alafenamide) or TDF (tenofovir disoproxil fumarate) and an Integrase inhibitor (dolutegravir)
  Interventions: Drug: Tenofovir; Drug: Dolutegravir

INTERVENTIONS:
Drug: Tenofovir — TAF (tenofovir alafenamide) or TDF(tenofovir disoproxil fumarate)
Drug: Rilpivirine — NNRTI
  Groups: Group A NRTI + NNRTI
Drug: Prezcobix — PI
  Groups: Group B NRTI + boosted PI
Drug: Dolutegravir — II
  Groups: Group C NRTI + II

SUMMARY:
This is a 3 arm, non-Interventional pilot single time point cross sectional study for the duration of 1 year. Total of 30 candidates (10 in each Group) will be enrolled into three different groups taking three different Antiretroviral regimen.

Based on current regimens that are commonly used (2017-2018 ART guidelines), our groups will include NRTI such as TAF (tenofovir alafenamide) or TDF(tenofovir disoproxil fumarate) plus one of the following:

Group A: an NNRTI (Non-nucleoside reverse transcriptase inhibitor, Rilpivirine Group B a boosted Protease Inhibitor: Prezcobix- [darunavir+cobicistat combination] Group C: an Integrase inhibitor (dolutegravir)

Once Informed Consent Process is obtained, blood will be drawn (55 ml) for stem/progenitor cell harvest and 15-20mls for biochemistry analysis. The Investigators will also obtain weight, waist-circumference, BP, pulse, BMI, Tanita body composition scale measures (which gives us body habitus measurements) and arterial stiffness measures.

DETAILED DESCRIPTION:
Metabolic and endocrine perturbations including insulin resistance, diabetes, and dyslipidemia have been of significant concern in human immunodeficiency virus (HIV)-infected individuals. HIV-infected individuals may be at risk of accelerated atherosclerotic cardiovascular disease (CVD) and metabolic syndrome. HIV infection itself and first-generation antiretroviral (ART) therapies, have been associated with adipose tissue/ lipodystrophic changes and disorders of glucose and lipid metabolism. More recent data suggest that immune activation and inflammation from chronic HIV infection may play an important role in HIV-associated metabolic dysfunction. Given the recent advances in ART, an increasing number of HIV-infected individuals are virologically controlled and living longer; as such, the trajectory of HIV-associated morbidity has shifted from one of primarily acute opportunistic infections and immune deficiency/dysfunction to one that includes chronic metabolic complications such as CVD. It is therefore important to discern the effect of current HIV medications on endothelial dysfunction and cardio-metabolic health.

Endothelial progenitor cells (EPCs), are an established biomarker for cardiovascular risk outcome measures. EPCs have been defined as CD34+ cells thereby identifying a defined homogenous population from heterogeneous peripheral blood derived mononuclear cells. We and others have previously shown that EPCs can act as a cellular biomarker that is more reliable than plasma-based markers for CVD risk estimation. Though these studies were not specifically directed towards HIV positive population one can postulate that CD34+ cells will act as an efficient biomarker for endothelial function in this population of interest.

Regarding treatment regimens for HIV, in general, the initial regimen for HIV-infected individuals usually includes two NRTIs plus an INSTI, an NNRTI, or a PI boosted with either cobicistat or ritonavir. Previously, protease inhibitors such as indinavir, and reverse transcriptase inhibitors such as AZT or d4t, have been implicated in mitochondrial dysfunction and oxidative stress, altered adipogenesis and differentiation, and impaired glucose and lipid homeostasis. Newer ART agents have been suggested to have lesser impact on metabolic parameters. However, these newer agents may trigger poorly understood processes that may have a negative impact on endothelium and numerous metabolic pathways.

Based on current regimens that are commonly used (2017-2018 ART guidelines), our groups will include NRTI such as TAF (tenofovir alafenamide) or TDF (tenofovir disoproxil fumarate) plus one of the following:

1: an NNRTI (Non-nucleoside reverse transcriptase inhibitor, Rilpivirine (Group A) 2. a boosted Protease Inhibitor: Prezcobix- [darunavir+cobicistat combination] (Group B), and 3: an Integrase inhibitor (dolutegravir) (Group C) We are including an integrase inhibitor because these agents have become the most popular initial regimen for newly infected HIV individuals. To avoid effect of medication within the three groups we have identified specific drugs within each class.

Significance: Although the etiology of metabolic/endocrine complications in HIV-infected individuals despite viremic control is poorly understood, it is most likely related to the interplay of host, viral, and ART factors and the complex interactions among the long-term consequences of infection, chronic ART, and the underlying inflammatory process. As mentioned before certain ARTs have raised concerns about metabolic dysfunction such as the PIs and it is important to determine whether other combination medications promote or reduce the chances of endothelial and metabolic dysregulation.

Pending a cure or vaccine to prevent HIV, a strong need exists to reduce long-term morbidity in HIV-infected individuals both by achieving viral suppression and limiting HIV- and/or ART-related complications, particularly since the current World Health Organization's guidelines recommend treating all HIV-infected individuals with ART. ) To discern endothelial function whole blood mononuclear cell derived EPC study is very appropriate. The Investigator have demonstrated that gene expression in EPCs change within two weeks of an intervention such as aerobic exercise. On the other-hand serum biomarkers usually take much longer time to change secondary to an intervention. The paracrine effect of damaged endothelium is secondary to gene expression changes that have been altered in the progenitor cells several months ahead of discernable changes in serum based biomarkers such as endothelium based inflammatory markers. When serum inflammatory markers are elevated that suggests that the endothelium is already damaged/ inflamed, possibly irreversibly.

EPCs are the future endothelium, therefore studying EPCs helps the Investigators to predict the effect of an intervention (such as a medication or exercise) on the future of endothelium and endothelial function. Their prime function is to migrate in response to a chemotactic factor such as SDF1 alpha, in order to repair the damaged or dysfunctional endothelium. In the normal course of events, EPCs transition to mature endothelium and replace endothelial cells after normal cell death cycle or programmed apoptosis. Unfortunately, obesity and HIV, both being pro-inflammatory, high reactive oxygen species (ROS) disease processes, chronically depletes the EPC population by up-regulating apoptotic pathways mediated by p53.

In order to understand the cellular mechanism(s) of chronic metabolic dysfunction and associated endothelial dysfunction leading to cardiovascular disease risk, in patients with HIV, it will be useful to study the peripheral blood derived endothelial progenitor cells (EPC, CD34+ cells) along with biochemistry, on three different treatment regimens and establish their effects on endothelium.

The Investigators believe this study design allows to discern whether the medication regimens have an effect on endothelium and biochemical parameters such as insulin, glucose, HbA1c, fasting lipid profile and also appetite controlling hormones. The latter has been particularly in focus lately with several diabetes medications, such as the incretins which modify appetite management pathway to treat obesity, metabolic syndrome, diabetes and reduce cardiovascular disease risk.

The arterial stiffness measure is a non-invasive procedure which provides the Investigators with important data on endothelial function and vascular health. Increased arterial stiffness indicates presence of increased peripheral resistance and predicts development of overt systolic and diastolic hypertension.

It is expected that EPC function studies would bear a negative correlation with biochemistry and arterial stiffness as demonstrated in other clinical trials. The biochemistry and arterial stiffness data as secondary outcome measure would help validate results and conclusions obtained from the primary outcome measures.

All together the Investigators have designed a study on HIV medication looking at their effect on endothelial function that is largely non-invasive yet giving valuable information on endothelial health, metabolic parameters and arterial stiffness. The study population is HIV positive patients, 40-70 years, male subjects only (to avoid gender differences during EPC based analysis), with a HbA1C less than 6.5% (subjects with no known history of diabetes). The study team will enroll 10 subjects from each group (A,B,C) who have been on a stable HIV regimen for at least one year. Total enrollment: 30 patients.

Innovation: This is an innovative study looking at different components of cardio-metabolic disease in HIV subjects and the role that HIV medication regimens play. The NIH is interested in this topic and has a current RFA out on this topic indicating lack of information. Our study design is unique as it combines cellular, biochemical and bio-physical components as outcome measures.

RESEARCH HYPOTHESIS The Investigators hypothesize that among these HIV regimens (A, B or C) there will be differences in the degree of metabolic derangement and endothelial dysfunction. The team plans to undertake a cross sectional study on HIV subjects on A, B or C regimens for at least one year, without diabetes, with known cardio-metabolic disease predisposition such as overweight and mild to moderate obesity (BMI 25.0- 39.9), but with no established coronary or cerebrovascular event

ELIGIBILITY:
Inclusion Criteria:

1. Male only (as gender variation of progenitor cells along with effect of estrogen, may lead to difficulty in data interpretation), Age above 40, but less than 70 years,
2. Body Mass Index (BMI) between 25.0-39.9 (both inclusive)
3. eGFR ≥ 50 mL/min/1.73 m2 by MDRD.

Exclusion Criteria:

1. Uncontrolled hyperglycemia with random blood glucose >200 mg/dL (>13.3 mmol/L)
2. Liver disease with ALT, AST or ALP x3 ULN
3. Subjects with HCV and HBV and detectable HCV RNA or HBV DNA
4. GFR <50 mL/min/1.73 m2 by MDRD
5. Prior surgery with chronic malabsorption (eg, bariatric) in prior 1 year
6. Clinically significant RBC disorders such as hemoglobinopathies
7. Chronic use of anti-inflammatory drugs for the last 3 months
8. On statin medications (ASCVD score less than or equal to 7.5%)
9. Use of consistent long-term steroid medication (oral, inhaled, injected) in last 1 month
10. Treatment with a strong cytochrome P450 3A4 (CYP34A) or P-gp inducer (ie:Rifampin)
11. Active smokers, Active wounds or recent surgery within 1 month
12. Untreated hyper/hypothyroidism
13. Implanted devices (eg. Pacemaker) that may interact with Tanita scale
14. Any other clinical condition that would jeopardize patient safety while participating
15. Women who are pregnant or breastfeeding
16. Chronic or persistent alcohol or drug abuse
17. Hypertriglyceridemia above 500mg/dl.
18. Prisoners or subjects who are involuntarily incarcerated
19. Subjects who are compulsorily detained for treatment of either a psychiatric illness
20. Participation in another trial with an investigational drug within 30 days prior to consent

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males from 40-70, with a Diagnosis of HIV, currently on HAART.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
CD34+/ total MNC percentage | Week 0, Single Time Point
  Percent of CD34+ cells over total Mononuclear cell
Colony Formation Capacity - Numbers of Colony formed | Week 0, Single Time Point
Migratory function in response to SDF1α | Week 0, Single Time Point
  How much the CD34+ cells migrate in response to SDF1a
Targeted gene expression of EPCs | Week 0, Single Time Point
  Gene expression

SECONDARY OUTCOMES:
Concentration of Serum Insulin | Week 0, Single Time Point
  to assess insulin resistance
Lipid Profile | Week 0, Single Time Point
  Cholesterol, LDL, HDL and TAG
Concentration Serum Leptin | Week 0, Single Time Point
  appetite controlling hormone
Arterial Stiffness through measuring Pulse wave Velocity | Week 0, Single Time Point
  through Pulse velocity

CONTACTS AND LOCATIONS:
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elzarki AF, Nandula SR, Awal H, Simon GL, Sen S. Cardiovascular disease (CVD) risk assessment of HIV medication regimens using hematopoietic CD34+ progenitor cells. Stem Cell Res Ther. 2022 Mar 7;13(1):103. doi: 10.1186/s13287-022-02775-6. PMID 35255964